CLINICAL TRIAL: NCT03845231
Title: Mucosal Correlates of Protection After Influenza Viral Challenge of Vaccinated and Unvaccinated Healthy Volunteers
Brief Title: Mucosal and Systemic Immunity After Viral Challenge of Healthy Volunteers Vaccinated With Inactivated Influenza Vaccine Via the Intranasal Versus Intramuscular Route
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 190058; 19-I-0058
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11-06

CONDITIONS: Influenza
Keywords: Human Challenge; Vaccine; Immune Response; Challenge Study; Healthy Volunteer
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- unvaccinated (Other): will receive no Flucelvax vaccination and will receive human challenge virus
  Interventions: Other: Human Challenge virus
- Vaccinated (Experimental): will receive Flucelvax vaccination and human challenge virus
  Interventions: Biological: Flucelvax(R); Other: Human Challenge virus

INTERVENTIONS:
Biological: Flucelvax(R) — Cohort 1 will receive IM quadrivalent IIV (Flucelvax (R)) at the standard dose of 15 micrograms HA per strain (60 micrograms HA total).
  Arms: Vaccinated
Other: Human Challenge virus — A dose of 10^7 50% tissue culture infective dose (TCID50) of human challenge virus will be administered intranasally to all participants using a nasal sprayer.

SUMMARY:
Background:

Influenza (flu) is a contagious respiratory virus that makes humans sick. Usually its symptoms are mild, but they can be dangerous. Researchers want to see if one way of giving the flu vaccine is more effective than another.

Objective:

To compare the body s ability to fight infection when a flu vaccine is given in the nose versus the arm.

Eligibility:

Healthy, nonsmoking adults ages 18 55. They must be willing to stay in isolation for at least 9 days. They must not have had the flu vaccine since September 1, 2018.

Design:

Participants must be willing to use birth control or abstinence from visit 1 until 8 weeks after getting the flu virus.

Participants will have at least 3 clinic visits over about a month. Visits may include:

Medical history

Physical exam

Blood and urine tests

Nasal samples collected

Heart and lung function tests

At the first visit, participants will get either:

Flu vaccine as injection in an arm muscle plus salt water sprays in the nose

OR flu vaccine as sprays in the nose plus salt water injection in an arm

Within the next few months, participants will stay in an isolation room for at least 9 days. They will be with up to 20 participants. Those who test positive for recreational drugs will leave the study. Participants will:

Repeat study tests

Answer questions about flu symptoms

Have the flu virus sprayed into their nose once

Be monitored by a medical team

Participants will have at least 2 follow-up visits and repeat study tests.

DETAILED DESCRIPTION:
The high morbidity and mortality associated with both pandemic and seasonal influenza and the threat of new potentially pandemic strains emerging makes influenza an important infectious disease and public health problem. Public health agencies must continue attempts to reduce the public health impact of this important virus.

Currently, influenza vaccination is the cornerstone of prophylaxis and the most effective method available to reduce the impact of influenza on the population. Current vaccines target the major surface protein, hemagglutinin (HA), and are standardized by stimulation of serum anti-HA antibodies as the primary correlate of protection. Measurements of serum antibodies to HA have become the gold standard for evaluating vaccines. The Food and Drug Administration (FDA) and the European Medicines Agency (EMA) Committee for Medicinal Products for Human Use (CHMP) both define protective titers as a hemagglutination inhibition (HAI) titer of greater than or equal to 40. Recent vaccine effectiveness has been limited and, in some populations, estimated at as low as 10%. Improved methods of vaccination must be developed, but limited information regarding the true correlates of protection is available. Correlates of protection in the systemic circulation may be less informative than those located in the nasopharyngeal mucosa, which is the site of exposure to and infection with influenza virus.

This study is designed to characterize the mucosal and systemic immunologic correlates of protection from influenza infection in persons vaccinated and unvaccinated against influenza. Half of participants will receive current licensed quadrivalent inactivated influenza vaccine (IIV) administered via the intramuscular (IM) route at the standard dose, prior to challenge with influenza virus. The other half will receive no vaccination prior to challenge. Immunologic response and clinical outcomes in the human challenge model will be determined to characterize the two cohorts. In the vaccinated cohort, mucosal and systemic immune responses induced by IM administration of quadrivalent IIV will also be carefully explored. The thoughtful study of mucosal immunity to influenza is expected to identify novel correlates of protection. By administering quadrivalent IIV and then infecting participants with human challenge virus, we can evaluate in detail the immunologic responses after immunization and subsequent virus exposure. This controlled setting offers the ideal environment to query these responses and to identify targets of mucosal stimulation for future vaccine strategies. In addition, the detailed characterization of the mucosal and systemic immune responses after vaccination and challenge will represent a true advance in understanding influenza immunity.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Greater than or equal to 18 and less than or equal to 55 years of age.
  2. Non-smoker.
  3. Have not received influenza vaccination of any type (whether licensed or unlicensed experimental vaccine) on or after September 1, 2018. Participants who enroll in our study must be informed of the Centers for Disease Control and Prevention (CDC) recommendation to receive seasonal influenza vaccination annually. Enrollees accept that half of study participants will receive licensed approved vaccination per the usual route, and half will receive it by an unapproved route with unknown efficacy and side effects. Enrollees should not plan to receive seasonal influenza vaccination from another source from enrollment through the final study visit (Phase 2, Day 56).
  4. Willingness to remain in isolation for the duration of viral shedding (at a minimum 9 days) and to comply with all study requirements.
  5. A male subject is eligible for the study if he meets one of the following criteria, beginning at least 4 weeks prior to enrollment and continuing until 8 weeks after administration of the human challenge virus:

     1. Is infertile, including history of successful vasectomy.
     2. Agrees to practice abstinence.
     3. Agrees that, with heterosexual intercourse with a fertile female partner, he will use a condom with spermicide and his female partner (including those who have undergone bilateral tubal ligation) will use an acceptable form of contraception (see inclusion criterion 6c).
  6. A female participant is eligible for this study if she is not pregnant or breastfeeding and meets one of the following criteria, beginning at least 4 weeks prior to enrollment and continuing until 8 weeks after administration of the human challenge virus::

     1. infertile, including postmenopausal status, (as defined by no menses for greater than or equal to 1 year) or history of hysterectomy.
     2. Agrees to practice abstinence.
     3. Agrees that, with heterosexual intercourse with a fertile male partner, she will use an acceptable form of contraception and her male partner will use a condom with spermicide. Acceptable effective methods of female contraception include the following: bilateral tubal ligation, implant of levonorgestrel, injectable progestogen, intrauterine device oral contraceptive pills and diaphragm with spermicide.
  7. Willing to have samples stored for future research.
  8. HIV uninfected with a negative test within 60 days of Phase 2, Day 0.
  9. Agrees not to use IN medications (including but not limited to nasal

     sprays, sinus rinses), over-the-counter medications (including but not

     limited to aspirin, decongestants, antihistamines, and other non-steroidal anti-inflammatory drugs), and herbal medications (including but not limited to herbal tea or St. John s Wort), from 14 days prior to study enrollment through the final study visit (Phase 2, Day 56), unless approved by the investigator
  10. Agrees not to donate blood or blood products from enrollment through the final study visit (Phase 2, Day 56).

EXCLUSION CRITERIA:

1. Presence of self-reported or medically documented significant medical condition including but not limited to:

   1. Chronic pulmonary disease (e.g., asthma, emphysema).
   2. Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
   3. Chronic medical conditions requiring close medical follow-up or hospitalization during the past 5 years (e.g., insulin-dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
   4. Immunosuppression, immune deficiency (such as IgA deficiency) or ongoing malignancy.
   5. Neurological and neurodevelopmental conditions (e.g., Bell s palsy, cerebral palsy, epilepsy, stroke, seizures).
   6. Postinfectious or postvaccine neurological sequelae including Guillain Barre syndrome.
   7. Individual with body mass index less than or equal to 18 and greater than or equal to 40.
2. Have close or household (i.e., share the same apartment or house) high-risk contacts including but not limited to:

   1. Persons greater than or equal to 65 years of age.
   2. Children less than or equal to 5 years of age.
   3. Residents of nursing homes.
   4. Persons of any age with significant chronic medical conditions such as:

      * Chronic pulmonary disease (e.g., severe asthma, chronic obstructive pulmonary disease).
      * Chronic cardiovascular disease (e.g., cardiomyopathy, congestive heart failure, cardiac surgery, ischemic heart disease, known anatomic defects).
      * Contacts who required medical follow-up or hospitalization during the past 5 years because of chronic metabolic disease (e.g., insulin-dependent diabetes mellitus, renal dysfunction, hemoglobinopathies).
      * Immunosuppression or cancer.
      * Neurological and neurodevelopmental conditions (e.g., cerebral palsy, epilepsy, stroke, seizures).
      * Individuals who are receiving long-term aspirin therapy.
      * Women who are pregnant or who are trying to become pregnant.
3. Acute illness within 7 days prior to quadrivalent IIV administration or inoculation with the human challenge virus.
4. Individuals who have grade 3 or above clinically significant laboratory values outside the limits thus specified by normal laboratory parameters.
5. Clinically significant abnormality as deemed by the PI on echocardiographic (ECHO) testing.
6. Clinically significant abnormality as deemed by the PI on the pulmonary function test (PFT).
7. Known allergy to influenza vaccination or excipients contained in the influenza vaccine used.
8. Known allergy to lidocaine or phenylephrine.
9. Known allergy to treatments for influenza (including but not limited to oseltamivir or nonsteroidal anti-inflammatory medications).
10. Known allergy to 2 or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
11. Anatomic or functional defects of the nasopharynx that could affect nasal sampling such as chronic rhinitis, nasal septal defect, nasal polyps or recent or remote nasal surgery
12. Receipt of blood or blood products (including immunoglobulins) within 3 months prior to enrollment.
13. Donation of blood or blood products within 3 months prior to study enrollment.
14. Receipt of any unlicensed drug within 3 months or 5.5 half-lives (whichever is greater) prior to enrollment.
15. Receipt of any unlicensed vaccine within 6 months prior to enrollment.
16. Self-reported or known history of alcoholism or drug abuse within 6 months prior to enrollment, or positive urine test for drugs of abuse (i.e., amphetamines, cocaine, benzodiazepines, opiates, metabolites, or tetrahydrocannabinol) at time of admission for viral challenge.
17. Self-reported or known history of psychiatric or psychological issues that require treatment and are deemed by the PI to be a contraindication to protocol participation.
18. Any condition or event that, in the judgment of the PI, is a contraindication to protocol participation or impairs the participant s ability to give informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Influenza infection | 1 yr
  The main focus of the study will be to characterize the mucosal and systemic immunologic correlates of protection from influenza infection in each of the two cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Memoli, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ainai A, Tamura S, Suzuki T, Ito R, Asanuma H, Tanimoto T, Gomi Y, Manabe S, Ishikawa T, Okuno Y, Odagiri T, Tashiro M, Sata T, Kurata T, Hasegawa H. Characterization of neutralizing antibodies in adults after intranasal vaccination with an inactivated influenza vaccine. J Med Virol. 2012 Feb;84(2):336-44. doi: 10.1002/jmv.22273. PMID 22170556
- [Background] Gould VMW, Francis JN, Anderson KJ, Georges B, Cope AV, Tregoning JS. Nasal IgA Provides Protection against Human Influenza Challenge in Volunteers with Low Serum Influenza Antibody Titre. Front Microbiol. 2017 May 17;8:900. doi: 10.3389/fmicb.2017.00900. eCollection 2017. PMID 28567036
- [Background] Flannery B, Chung JR, Belongia EA, McLean HQ, Gaglani M, Murthy K, Zimmerman RK, Nowalk MP, Jackson ML, Jackson LA, Monto AS, Martin ET, Foust A, Sessions W, Berman L, Barnes JR, Spencer S, Fry AM. Interim Estimates of 2017-18 Seasonal Influenza Vaccine Effectiveness - United States, February 2018. MMWR Morb Mortal Wkly Rep. 2018 Feb 16;67(6):180-185. doi: 10.15585/mmwr.mm6706a2. PMID 29447141
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-I-0058.html